CLINICAL TRIAL: NCT00879047
Title: Interaction of Alcohol & HAART in HIV/AIDS and HIV/AIDS With HCV Co-Infection
Brief Title: Interaction of Alcohol and Highly Active Antiretroviral Therapy (HAART) in HIV/AIDS and HIV/AIDS With Hepatitis C Virus (HCV) Co-Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double
Other Study IDs: R01AA018001 (NIH)
Record Dates: First submitted 2009-03-24; First posted 2009-04-09 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: HIV Infections; Hepatitis C
Keywords: HIV; Hepatitis C
MeSH Terms: conditions — HIV Infections; Hepatitis C | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- HIV+, Ritonavir-regimen (Experimental): 10 subjects will be HIV+ and will begin receiving Ritonavir-containing regimen, and their PK interactions with alcohol/placebo will be evaluated.
  Interventions: Drug: Alcohol; Drug: Alcohol placebo
- HIV+/HCV+ Co-infected, Ritonavir-regimen (Experimental): 10 subjects will be HIV+/HCV+ co-infected and will begin receiving Ritonavir-containing regimen, and their PK interactions with alcohol/placebo will be evaluated.
  Interventions: Drug: Alcohol; Drug: Alcohol placebo
- HIV+, Efavirenz-regimen (Experimental): 10 subjects will be HIV+ and will begin receiving Efavirenz-containing regimen, and their PK interactions with alcohol/placebo will be evaluated.
  Interventions: Drug: Alcohol; Drug: Alcohol placebo
- HIV+/HCV+ Co-infected, Efavirenz-regimen (Experimental): 10 subjects will be HIV+/HCV+ co-infected and will begin receiving Efavirenz-containing regimen, and their PK interactions with alcohol/placebo will be evaluated.
  Interventions: Drug: Alcohol; Drug: Alcohol placebo
- Maraviroc in Healthy Subjects (Experimental): 10 healthy subjects will begin receiving maraviroc, and their PK interactions with alcohol/placebo will be evaluated.
  Interventions: Drug: Alcohol; Drug: Alcohol placebo

INTERVENTIONS:
Drug: Alcohol — Consumed orally as liquid mixed with a juice beverage, 1 g/kg formula, administered once at baseline and again at either 2 or 3 weeks
  Other Names: grain alcohol
Drug: Alcohol placebo — Liquid alcohol spritzed on top of juice beverage immediately prior to administration in order to give smell of alcohol, administered once at baseline and again at either 2 or 3 weeks
  Other Names: grain alcohol

SUMMARY:
The proposed studies will examine the extent of pharmacokinetic and pharmacodynamic interactions between alcohol and various antiretroviral therapies in those with HIV/AIDS, HIV/HCV co-infection, mild HCV and healthy subjects.

DETAILED DESCRIPTION:
The goal of this research study is to improve the clinical care of human immunodeficiency virus (HIV)-infected or HIV/Hepatitis C (HCV) co-infected, alcohol-using patients by identifying significant interactions which may occur between drugs commonly used to treat HIV disease known to be cytochrome P450 (CYP450) inducers or inhibitors and alcohol, the most frequently abused substance in the United States. We hypothesize that concomitant use of alcohol and currently utilized antiretroviral therapy (ART) will be associated with significant drug interactions including alteration of alcohol and ART pharmacokinetics as well as altered responses to alcohol administration. We plan to conduct alcohol and ART administration studies in 6 study samples (n=10 each): 1. those with HIV/AIDS and eligible for efavirenz-containing HAART, 2. those with HIV/AIDS and eligible for a ritonavir-boosted protease inhibitor based HAART, 3. those with HIV/AIDS and HCV eligible for an efavirenz-containing HAART, 4. those with HIV/AIDS and HCV eligible for a ritonavir-boosted protease inhibitor regimen, 5. healthy subjects taking clinically relevant doses of maraviroc and 6. those with mild HCV taking clinically relevant doses of maraviroc. Pharmacokinetics, subjective, and cognitive data will be serially collected over the course of study sessions where either alcohol or placebo is administered prior to and following ART. Data collected will elucidate the presence and clinical significance of drug interactions, both pharmacokinetic and pharmacodynamic, between alcohol and ART in these populations.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be diagnosed with HIV/AIDS, HIV/AIDS and Hepatitis C, mild Hepatitis C or will be healthy as determined by history and physical examination, screening laboratory tests and urinalysis, and will be eligible for treatment with HAART
* Participants will be experienced with alcohol consumption
* They may meet diagnostic criteria for alcohol abuse or non-physiological alcohol dependence, but may not be dependent on any other substances including opioids, stimulants, cannabis, hallucinogens or other substances, prescribed or illicit
* For those with HCV coinfection, HCV must be at a stage consistent with no more than mild liver fibrosis (fibrosis stage assessed by two methods: the AST to platelet ratio (APRI) (at a score of <0.5 for eligibility) and the FIB-4 fibrosis index (score of <1.5 for eligibility), both of which indicate mild liver disease.)
* Age 21 or older
* Hemoglobin Men > 11 g/dL, Women > 10 g/dL5
* Able to give voluntary, signed, informed consent.

Exclusion Criteria:

* Patients who are receiving concurrently other drugs that are inducers or inhibitors of hepatic microsomal enzymes
* Patients with a known sensitivity to the HIV therapeutics to be studied
* Pregnant women or nursing mothers.
* All women who are sexually active and capable of becoming pregnant must have a negative pregnancy test within one week prior to entry into these studies.
* Major psychotic illness or suicidality.
* Clinically active hepatitis with liver enzyme elevations > 3 times the upper limit of normal or evidence of liver fibrosis at a stage indicative of greater than mild stage for fibrosis (see Inclusion Criteria).
* Those with obesity (BMI > 30), diabetes, hyperlipidemia, coagulation disorders, or renal disease will be excluded.
* Hemoglobin Men < 11 g/dL, Women < 10 g/dL
* Physical dependence on alcohol.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Plasma levels of antiretroviral medications. | Baseline, two weeks, and three weeks.
Plasma levels of alcohol. | Baseline, two weeks, and three weeks.

SECONDARY OUTCOMES:
Measures of cognitive and behavioral change/impairment. | Baseline, two weeks, and three weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Elinore F McCance-Katz, M.D., Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States